CLINICAL TRIAL: NCT06391762
Title: Level of Deprivation Assessment in the Population of Short-bowel Syndrome With Intestinal Failure Patients Monitored by the Nancy University Hospital, France, Between 2020 and 2023
Brief Title: Level of Deprivation Assessment in a Population of Short-bowel Syndrome Patients With Intestinal Failure
Acronym: PRECAR-SGC
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, MICHOT Niasha, Principal Investigator, Central Hospital, Nancy, France
Other Study IDs: 2023PI056
Record Dates: First submitted 2024-04-22; First posted 2024-04-30 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Short Bowel Syndrome; Intestinal Failure; Deprivation, Psychosocial
MeSH Terms: conditions — Short Bowel Syndrome; Intestinal Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The association between social deprivation and chronic disease is regularly examined but there are no data available on patients with intestinal failure due to short bowel syndrome (SBS-IF). First, the investigators aim to characterize this population and then to assess if insecurity is associated with some disease criteria.

DETAILED DESCRIPTION:
This exploratory cross-sectional study was conducted on patients affected by intestinal failure in short bowel syndrome and monitored by the certified home parenteral nutrition (HPN) center of Nancy University Hospital.

The investigators included all patients over 18 years old suffering from SBS-IF followed-up by the certified HPN center of Nancy University Hospital between March 1st, 2020, and November 30th, 2023.

The f-EDI (a European ecological index adapted to France) was determined for each participant.

The investigators set the initial date at 2020, as this corresponds to the start of the use of patient-specific formulas in the center. Exclusion criteria were: not living in France, because it's required to use French-EDI and patients under 18 years old because they are monitored by the children's hospital. Investigators also excluded patients with transitory type 1 SBS who would have a bowel length over 2 meters after re-establishment of digestive continuity.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age
* Suffering from Short-bowel syndrome with intestinal failure
* Monitored by the Certified Home Parenteral Nutrition Center of the Nancy University Hospital
* Between March 1st 2020 and November 30th 2023

Exclusion Criteria:

* Patients not living in France
* Transitory short-bowel syndrome with a predicted bowel length > 200cm after digestive continuity

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients over 18 years of age suffering from Short-bowel syndrome with intestinal failure, monitored by the Certified Home Parenteral Nutrition Center of the Nancy University Hospital, between March 1st 2020 and November 30th 2023
Sampling Method: Non-Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2023-12-28 (Actual); Primary Completion 2024-01-03 (Actual); Study Completion 2024-01-03 (Actual)

PRIMARY OUTCOMES:
Deprivation level | Throughout study completion, an average of 1 month
  Determine the deprivation level of this population using the f-EDI of each participant

SECONDARY OUTCOMES:
Association between deprivation level and disease characteristics | Throughout study completion, an average of 1 month
  Determine the association between the deprivation level of the patients with SBS-IF determined by f-EDI and the characteristics of their disease

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU Nancy, Vandœuvre-lès-Nancy, Lorraine, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tudrej BV, Martinière A, Etonno R, et al. Scores de précarité en pratique clinique. Médecine. 2019;15(3):117-125
- [Background] Merville O, Launay L, Dejardin O, Rollet Q, Bryere J, Guillaume E, Launoy G. Can an Ecological Index of Deprivation Be Used at the Country Level? The Case of the French Version of the European Deprivation Index (F-EDI). Int J Environ Res Public Health. 2022 Feb 17;19(4):2311. doi: 10.3390/ijerph19042311. PMID 35206501
- [Background] Pironi L, Boeykens K, Bozzetti F, Joly F, Klek S, Lal S, Lichota M, Muhlebach S, Van Gossum A, Wanten G, Wheatley C, Bischoff SC. ESPEN practical guideline: Home parenteral nutrition. Clin Nutr. 2023 Mar;42(3):411-430. doi: 10.1016/j.clnu.2022.12.003. Epub 2023 Jan 9. PMID 36796121
- [Background] Pironi L. Definitions of intestinal failure and the short bowel syndrome. Best Pract Res Clin Gastroenterol. 2016 Apr;30(2):173-85. doi: 10.1016/j.bpg.2016.02.011. Epub 2016 Feb 18. PMID 27086884
- [Background] Pironi L, Steiger E, Joly F, Jeppesen PB, Wanten G, Sasdelli AS, Chambrier C, Aimasso U, Mundi MS, Szczepanek K, Jukes A, Theilla M, Kunecki M, Daniels J, Serlie M, Poullenot F, Cooper SC, Rasmussen HH, Compher C, Seguy D, Crivelli A, Santarpia L, Guglielmi FW, Kozjek NR, Schneider SM, Ellegard L, Thibault R, Matras P, Matysiak K, Van Gossum A, Forbes A, Wyer N, Taus M, Virgili NM, O'Callaghan M, Chapman B, Osland E, Cuerda C, Udvarhelyi G, Jones L, Won Lee AD, Masconale L, Orlandoni P, Spaggiari C, Diez MB, Doitchinova-Simeonova M, Serralde-Zuniga AE, Olveira G, Krznaric Z, Czako L, Kekstas G, Sanz-Paris A, Jauregui MEP, Murillo AZ, Schafer E, Arends J, Suarez-Llanos JP, Youssef NN, Brillanti G, Nardi E, Lal S; Home Artificial Nutrition and Chronic Intestinal Failure Special Interest Group of ESPEN; European Society for Clinical Nutrition and Metabolism. Characteristics of adult patients with chronic intestinal failure due to short bowel syndrome: An international multicenter survey. Clin Nutr ESPEN. 2021 Oct;45:433-441. doi: 10.1016/j.clnesp.2021.07.004. Epub 2021 Jul 28. PMID 34620351
- [Background] Calvar E, Launay L, Boyer A, Launoy G, Lobbedez T, Chatelet V. Effects of Social Deprivation on the Proportion of Preemptive Kidney Transplantation: A Mediation Analysis. Transplant Direct. 2021 Sep 7;7(10):e750. doi: 10.1097/TXD.0000000000001203. eCollection 2021 Oct. PMID 36567853
- [Background] Winkler MF, Smith CE. Clinical, social, and economic impacts of home parenteral nutrition dependence in short bowel syndrome. JPEN J Parenter Enteral Nutr. 2014 May;38(1 Suppl):32S-37S. doi: 10.1177/0148607113517717. Epub 2014 Jan 13. PMID 24418898